CLINICAL TRIAL: NCT03511404
Title: Clinical Electrophysiology Assessment for Rehabilitation Progress of Low Back Pain Patients
Brief Title: Clinical Electrophysiology Assessment for Low Back Pain
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong HU, Associate Professor, The University of Hong Kong
Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0132
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Non Specific Chronic Low Back Pain
Keywords: Non specific chronic low back pain; surface electromyography (EMG); neuromuscular function; physiotherapy; Numeric Pain Rating Scale

STUDY DESIGN:
Intervention Model Description: A correlation study between clinical examination by Numeric Pain Rating Scale (NPRS) and electrophysiology assessment by surface EMG will be conducted at enrollment and 6 weeks physiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronical LBP (Experimental): Patients with chronic low back pain to be measured with Numeric Pain Rating Scale (NPRS).
  Interventions: Other: physiotherapy rehabilitation

INTERVENTIONS:
Other: physiotherapy rehabilitation — All subjects will receive a course of conventional physiotherapy that incorporating components of pain relief and functional restoration with the use of electrotherapy and exercise therapy for twelve sessions twice weekly in six weeks guided by a registered physiotherapist in Hong Kong.

SUMMARY:
Non specific chronic low back pain (LBP) is a debilitating disorder characterized by tremendous personal and socioeconomic impact, with long-term sick leave, low quality of life, and very high financial costs. Evidence suggests that patients with non specific LBP presented with altered muscle activity pattern when compare with healthy people. It has been reviewed that exercise therapy was effective for modulation of muscle dysfunction in chronic low back pain. However, there is a lack of objective assessment of the pain relief in low back pain rehabilitation. Clinical application of surface electromyography (EMG) may provide a quantitative and objective tool to evaluate the rehabilitation outcome in patients with non specific chronic low back pain before and after treatment.

Objectives: To verify the usefulness of surface electromyography (EMG) in low back pain (LBP) rehabilitation assessment.

Setting: Out-patient physiotherapy musculoskeletal rehabilitation

DETAILED DESCRIPTION:
Participants: One hundred adults with non specific chronic low back pain (LBP) will be recruited.

Methodology: A prospective correlation study between clinical examination and electrophysiology assessment. This project will perform carefully with a definitive chronic low back pain (LBP). Firstly, we will compare the surface EMG features from patients with LBP to normal data. In addition, the changes in electrophysiology assessment will be compared with clinical assessment by Numeric Pain Rating Scale (NPRS). This allows us to verify the potential clinical application of surface EMG features in physiotherapy progress assessment.

ELIGIBILITY:
Inclusion Criteria:

* One hundred persons with non specific low back pain will be recruited consecutively from the Specialist Outpatient Department (SOPD) of Physiotherapy Department of Queen Elizabeth Hospital. Subjects will be included in the study if they presented with symptom duration of greater than three months with no radiological abnormality detected.

Exclusion Criteria:

* All subjects should be able to provide informed consent and demonstrate sufficient ability to tolerate the experiment procedure to avoid aggravation of symptoms during the experiment procedures. Subjects will be excluded if they have any major orthopedic, neurological, circulatory or respiratory conditions, a history or family history of epilepsy, recent or current pregnancies, and previous surgery to the abdomen or back. The back pain history in the previous year will be documented for those eligible subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline on enrollment and after six weeks physiotherapy
  Intensity of self-reported pain was measured using a Numeric Pain Rating Scale (NPRS) anchored with 'no pain' at 0 and 'worst pain imaginable' at 10. Subjects rated their average pain over the preceding month prior to motor training, and rated their average pain across the final week of motor training.

SECONDARY OUTCOMES:
surface electromyography (EMG) | Baseline on enrollment and after six weeks physiotherapy
  Disposable surface EMG electrodes will be attached in array to the right and left lumbar erector spinae (LES) muscles, approximately 2 cm lateral to the L3 spinous process. Root mean square amplitude of surface EMG measured was calculated and flexion-relaxation ratio in sitting was formulated by dividing the average surface EMG activity in upright sitting by the average surface EMG activity in slumped sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- Electromyography (EMG)system, Zhuhai, Guangdong, China